CLINICAL TRIAL: NCT06269822
Title: Electrophysiological Evaluation of Autonomic Dysfunction in Persons With Temporal Lobe Epilepsy and Its Relation Ship With Sudden Unexpected Death of Epileptic Patient (SUDEP) Risk Development(
Brief Title: Autonomic Dysfunction in Temporal Lobe Epilepsy and SUDEP
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Reem Mahmoud Gabr, doctor, Cairo University
Other Study IDs: SSR, HRV, QEEG in TLE
Record Dates: First submitted 2024-02-10; First posted 2024-02-21 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2024-02

CONDITIONS: Temporal Lobe Epilepsy
Keywords: Temporal Lobe epilepsy (TLE); Sudden unexpected death of epileptic patients (SUDEP); Dysautonomia; Quantitative EEG (QEEG); Sympathetic Skin Response (SSR); Heart Rate Variability (HRV)
MeSH Terms: conditions — Epilepsy, Temporal Lobe; Autonomic Nervous System Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cases: Group-1: Patients with TLE of both genders and aged > 18 years old
  Interventions: Diagnostic Test: Sympathetic skin response, heart rate variability test, quantitative EEG
- Controls: Group-2: Age/gender matched healthy controls
  Interventions: Diagnostic Test: Sympathetic skin response, heart rate variability test, quantitative EEG

INTERVENTIONS:
Diagnostic Test: Sympathetic skin response, heart rate variability test, quantitative EEG — Sympathetic skin test (electrodermal activity) to test for sympathetic function Heart rate variability test to assess cardiovagal function Quantitative EEG to quantitatively assessing the brain function using fast fourier transform technique

SUMMARY:
The study aimed at detection of autonomic dysfunction among cases with temporal lobe epilepsy; using different electrophysiological techniques.

Moreover, it aimed at finding any correlation between electrophysiological tests and SUDEP risk.

DETAILED DESCRIPTION:
Temporal lobe epilepsy (TLE) is the commonest focal form of epilepsy; representing 60% of all epilepsies . It has two major subtypes; neocortical (nTLE) and mesial (mTLE), each with different presentations.

Its diagnosis depends on detailed clinical history, neurological examination as well as neurophysiological (including EEG), and neuroimaging diagnostic tests which are mandatory in localizing the pathology.

Intimate connection between epileptic networks and the autonomic nervous system had been revealed. Seizures could affect autonomic functions whether directly through activation of cortical autonomic centers or indirectly through the released catecholamines.

The SUDEP is considered as one of the most serious complications of epilepsy and second most common cause of death from neurological diseases after stroke. Autonomic dysfunction could have a potential role in the pathophysiology of sudden unexpected death of epileptic patients (SUDEP).

Attention has been focused on biomarkers that could assist in the detection and early stratification of SUDEP risk. Such biomarkers include neurophysiological tests, imaging findings, laboratory findings.

Among the introduced neurophysiological biomarkers are electroencephalogram (EEG), sympathetic skin response (SSR) and heart rate variability (HRV).

The HRV is considered as simple, sensitive index of cardiovagal function. Reduced heart rate variability (HRV) is a strong predictor of sudden death in patients with heart disease.

The electrodermal activity (EDA )or SSR is referred as the most popular used test for assessment the sudomotor function . The EDA had been proven to be a reliable biomarker for detecting generalized tonic-clonic seizures (GTCs) through a wearable device.

Frontal midline theta activity was studied using quantitative EEG (QEEG); that confirmed the presence of interactive relationships between activities of the peripheral autonomic system and the cortical network. The QEEG technique had been introduced in the thirties of the last century. Yet, it had not been applied before on epileptic patients to assess either the central autonomic function or the SUDEP risk and thus, this is considered as the first study to address such issue.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed as temporal lobe epilepsy(TLE) depending on clinical semiology and EEG temporal inter-ictal epileptiform discharges

Exclusion Criteria:

* Any identifiable disease that could affect autonomic nervous system function including diabetic patients.
* Any drug that could affect autonomic nervous system function including oral contraceptives

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Out-patient epilepsy clinic at kasr alainy hopsital -Cairo University
Sampling Method: Non-Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-11-25 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
Detection of autonomic dysfunction (sympathetic domain) among cases of temporal lobe epilepsy | 30 minutes was the estimated test time. Outcome was assessed through study completion
  Assessing the sympathetic domain of the autonomic nervous system using sympathetic skin response (SSR) test; in which response latency and amplitude were measured and then compared to the matched controls (higher amplitude signifying higher sympathetic tone)
Detection of autonomic dysfunction (Para-sympathetic domain) among cases of temporal lobe epilepsy | 20 minutes was the estimated test time. Outcome was assessed through study completion
  Evaluating the parasympathetic domain of the ANS using the heart rate variability test(HRV); in which root mean square of successive differences (RMSSD) as a time domain parameter was measured and then compared to the matched controls ( Reduced RMSSD denoting reduced vagal tone)

SECONDARY OUTCOMES:
Detection of the sudden unexpected death of epileptic patient (SUDEP) risk using Quantitative EEG (QEEG) in temporal lobe epilepsy(TLE) patients | 30-45 minutes is the estimated test time. Outcome was assessed through study completion
  Assessing of certain QEEG parameter could help in identifying patients with high SUDEP risk. SUDEP risk was evaluated using SUDEP-7 inventory score (7 questions each with 1 point); patients with higher score are assumed to have higher risk for developing sudden death.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Neurophysiology unit- Kasr alainy-Cairo University, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Clemens B, Emri M, Fekete I, Fekete K. Epileptic diathesis: An EEG-LORETA study. Clin Neurophysiol. 2023 Jan;145:54-61. doi: 10.1016/j.clinph.2022.11.004. Epub 2022 Nov 17. PMID 36442376
- [Background] Barot N, Nei M. Autonomic aspects of sudden unexpected death in epilepsy (SUDEP). Clin Auton Res. 2019 Apr;29(2):151-160. doi: 10.1007/s10286-018-0576-1. Epub 2018 Nov 19. PMID 30456432
- [Background] Vieluf S, El Atrache R, Hammond S, Touserkani FM, Loddenkemper T, Reinsberger C. Peripheral multimodal monitoring of ANS changes related to epilepsy. Epilepsy Behav. 2019 Jul;96:69-79. doi: 10.1016/j.yebeh.2019.02.018. Epub 2019 May 14. PMID 31100658